CLINICAL TRIAL: NCT06102408
Title: Relevance and Efficiency of SecOnd Line Workup for Uveitis
Acronym: RESOLVE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Thomas MOULINET, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2023PI190
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with only one etiological workup: patients who underwent only one set of exams for etiological investigations of uveitis
  Interventions: Other: second line investigations for uveitis etiological workup
- Patients without diagnostic modification subsequently to the second etiological workup: Patients who underwent a second etiological workup, independently of the results of the fist line investigations, and whose diagnosis was not modified by the second line investigations.
  Interventions: Other: second line investigations for uveitis etiological workup
- Patients with diagnostic modification subsequently to the second etiological workup: Patients who underwent a second etiological workup, independently of the results of the fist line investigations, and whose diagnosis was modified by the second line investigations.
  Interventions: Other: second line investigations for uveitis etiological workup

INTERVENTIONS:
Other: second line investigations for uveitis etiological workup — Biological, radiological or histological investigations performed after a first line etiological workup. Investigations conducted following abnormal resultats of first line exams were not considered as second line exams (e.g. : bronchoscopy performed after abrnomal CT scan).

SUMMARY:
The first-line etiological workup is currently poorly codified, and some patients undergo sequential investigations. However, the reason which lead the clinician to perform subsequent exams, and the relevance of such exams, remain to be determined. The main objective of the study was to assess the relevance of a second-line workup of patients with uveitis.

DETAILED DESCRIPTION:
The first-line etiological workup is currently poorly codified, with some patients undergoing extensive investigations, and other minimal etiological workup. In addition, some patients undergo sequential investigations. However, the reason which lead the clinician to perform subsequent exams, and the relevance of investigations performed after a first line workup remain to be determined. The main objective of the study was to assess the relevance of a second-line workup of patients with uveitis.Secondary objectives were to describe the reasons of these second-line workups, and to determine which exams were the most relevant, and the determinants of its realization.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* at least one etiological workup in our center

Exclusion Criteria:

* only episode of acute anterior uveitis quickly responding to topical treatments
* diagnostic ophthalmologically obvious
* opposition to collection of data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult pateints with uveitis requiring at least one etiological workup.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
patients undergoing a second line etiological workup | through study completion, an average of 18 months
  percentage of patients undergoing a second line etiological workup

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hwang DK, Chou YJ, Pu CY, Chou P. Epidemiology of uveitis among the Chinese population in Taiwan: a population-based study. Ophthalmology. 2012 Nov;119(11):2371-6. doi: 10.1016/j.ophtha.2012.05.026. Epub 2012 Jul 17. PMID 22809756
- [Background] Dandona L, Dandona R, John RK, McCarty CA, Rao GN. Population based assessment of uveitis in an urban population in southern India. Br J Ophthalmol. 2000 Jul;84(7):706-9. doi: 10.1136/bjo.84.7.706. PMID 10873978
- [Background] Jabs DA, Nussenblatt RB, Rosenbaum JT; Standardization of Uveitis Nomenclature (SUN) Working Group. Standardization of uveitis nomenclature for reporting clinical data. Results of the First International Workshop. Am J Ophthalmol. 2005 Sep;140(3):509-16. doi: 10.1016/j.ajo.2005.03.057. PMID 16196117
- [Background] Smith JR, Rosenbaum JT. Management of uveitis: a rheumatologic perspective. Arthritis Rheum. 2002 Feb;46(2):309-18. doi: 10.1002/art.503. No abstract available. PMID 11840433
- [Background] Selmi C. Diagnosis and classification of autoimmune uveitis. Autoimmun Rev. 2014 Apr-May;13(4-5):591-4. doi: 10.1016/j.autrev.2014.01.006. Epub 2014 Jan 12. PMID 24424168
- [Background] de Parisot A, Jamilloux Y, Kodjikian L, Errera MH, Sedira N, Heron E, Perard L, Cornut PL, Schneider C, Riviere S, Olle P, Pugnet G, Cathebras P, Manoli P, Bodaghi B, Saadoun D, Baillif S, Tieulie N, Andre M, Chiambaretta F, Bonin N, Bielefeld P, Bron A, Mouriaux F, Bienvenu B, Amamra N, Guerre P, Decullier E, Seve P; ULISSE group. Evaluating the cost-consequence of a standardized strategy for the etiological diagnosis of uveitis (ULISSE study). PLoS One. 2020 Feb 14;15(2):e0228918. doi: 10.1371/journal.pone.0228918. eCollection 2020. PMID 32059021